CLINICAL TRIAL: NCT02493023
Title: Assessment of a Novel, Fast and Automatic CT-to-patient Registration Method During Navigated Bronchoscopy and Endobronchial Ultrasound Bronchoscopy (EBUS)
Brief Title: Automatic CT-to-patient Registration During Navigated Bronchoscopy and EBUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/3385
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Bronchial Neoplasms
Keywords: Bronchoscopy; Bronchoscopes
MeSH Terms: conditions — Bronchial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- navigated bronchoscopy (Experimental)
  Interventions: Device: navigated bronchoscopy

INTERVENTIONS:
Device: navigated bronchoscopy
  Other Names: position tracked bronchoscope; navigated endobronchial ultrasound (EBUS)

SUMMARY:
Bronchoscopic diagnosis and staging of lung cancer must be gentle and quick, and requires optimal sampling precision.Electromagnetic navigation systems are promising for intraoperative guiding based on maps made of preoperative CT images. Navigation accuracy depends largely on correct alignment of preoperative images to the patient´s position in space during endoscopy. In this study, the accuracy of a new fast and automatic image-to-patient registration method during the initial phase of bronchoscopy is assessed in patients referred for lung cancer investigation.

DETAILED DESCRIPTION:
This is an accuracy study of a new automatic CT-to-patient registration technique for bronchoscopy and endobronchial ultrasound bronchoscopy (EBUS). An in-house research and development navigation platform displays the intraoperative position of the endoscope inside the airways, and shows its exact position in three-dimensional (3D) maps made from the patients' own preoperative CT images. The navigation system is used for acquiring position data from a bronchoscope or EBUS-scope (same sort of output data acquired from both endoscopes in this study) equipped with a position sensor for electromagnetic tracking. From intraoperative position data, the accuracy of the image-to-patient registration and the navigation system accuracy can be calculated. When targeting a certain lymph node or tumor for sampling, the pulmonologist can use electromagnetic navigation combined with preoperative CT images to navigate directly, precisely and accurately to the area of interest. Functional systems for navigated bronchoscopy and EBUS may therefore lead to considerable improvements in lung cancer diagnosis and mediastinal staging.

ELIGIBILITY:
Inclusion Criteria:

* referred to thoracic department St Olavs Hospital due to suspicion of lung cancer
* informed consent

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
endoscope position (measured in millimetres from origo in the x, y and z-plane) in 3 dimensional maps from preoperative CT images | 48 hours
  intraoperative positional data of bronchoscope or endobronchial ultrasound scope (EBUS) measured and stored in navigation system software, used for registration and navigation system accuracy calculations

SECONDARY OUTCOMES:
duration of procedure | 48 hours
  time from first entry of endoscope through vocal cords to final withdrawal of endoscope
patient reported satisfaction | 48 hours
  enquiry on patients´own experience 2 hours after end of navigated bronchoscopy/EBUS procedure
adverse events | 48 hours
  procedure related adverse events or unexpected incidents registrated

CONTACTS AND LOCATIONS:
Overall Officials: Toril A Nagelhus Hernes, prof, Study Director — Department of Circulation and Imaging
Locations (1):
- Department of Thoracic Medicine, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Sorger H, Hofstad EF, Amundsen T, Lango T, Leira HO. A novel platform for electromagnetic navigated ultrasound bronchoscopy (EBUS). Int J Comput Assist Radiol Surg. 2016 Aug;11(8):1431-43. doi: 10.1007/s11548-015-1326-7. Epub 2015 Nov 28. PMID 26615428